CLINICAL TRIAL: NCT05320978
Title: Association of Preoperative Sarcopenia and Intraoperative Hypotension in Patients Undergoing Minimally Invasive Pylorus Preserving Pancreaticoduodenectomy : Prospective Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2022-0135
Record Dates: First submitted 2022-04-03; First posted 2022-04-11 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Patients Undergoing Minimally Invasive Pylorus Preserving Pancreaticoduodenectomy
MeSH Terms: interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients undergoing minimally invasive pylor-preserving pancreaticoduodenectomy: Adult patients aged 20 years or older and who underg minimally invasive pylor-preserving pancreaticoduodenectomy
  Interventions: Device: Hand grip test, computed tomography

INTERVENTIONS:
Device: Hand grip test, computed tomography — A hand grip test, abdominal computed tomography are performed before surgery.

SUMMARY:
The aim of this study is to determine whether preoperative sarcopenia (low muscle strength/muscle mass) is correlated with time weighted average intraoperative hypotension in patients undergoing minimally invasive pylorus preserving pancreaticoduodenectomy.

ELIGIBILITY:
Inclusion Criteria:

1. patients 20 years or older who undergo minimally invasive pylorus preserving pancreaticoduodenectomy

Exclusion Criteria:

1. emergency surgery
2. patients who cannot read consent forms(e.g., illiterate, foreigner, etc.)
3. patients with cognitive dysfunction
4. pregnant, lactating women
5. When hand grip test cannot be performed
6. patients with atrial fibrillation, moderate or severe valvular heart disease, left ventricular ejection fraction less than 35%

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing minimally invasive pylorus preserving pancreaticoduodenectomy
Sampling Method: Non-Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2024-03-27 (Estimated); Study Completion 2024-03-27 (Estimated)

PRIMARY OUTCOMES:
time weighted average intraoperative hypotension | Procedure (From the induction of anesthesia to the end of anesthesia)
  1) Intraoperative hypotension is defined as a mean blood pressure < 65 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: So Yeon Kim, MD,PhD, Principal Investigator — Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Korea.
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided